CLINICAL TRIAL: NCT05976867
Title: Parent-focused Primary Prevention of Child Sexual Abuse: An Effectiveness-implementation Hybrid Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD108209 (NIH)
Record Dates: First submitted 2022-12-06; First posted 2023-08-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Child Sexual Abuse
Keywords: primary prevention; child sexual abuse; implementation science

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAT + Smart Parents (Experimental): Participants in this arm will receive the additional Smart Parents module, added to Parents as Teachers (PAT) in which they are already enrolled. This is the experimental condition.
  Interventions: Behavioral: Parents as Teachers (PAT) + Smart Parents
- PAT as usual (Active Comparator): Participants in this arm will continue to receive Parents as Teachers (PAT) as usual. This is the treatment as usual condition (comparison).
  Interventions: Behavioral: Parents as Teachers (PAT) as usual

INTERVENTIONS:
Behavioral: Parents as Teachers (PAT) as usual — Parents as Teachers parent-education program as designed. Delivered in the home to parents of children under 5. Parents begin with the foundational curriculum (mostly taught within the first six sessions) focused on healthy child development, parenting behaviors including parent-child interactions and communication, and creating a safe home environment in terms of avoiding accidents and injuries. After the foundational curriculum, additional sessions are delivered based on the continued needs of the family until the child ages out or the parent discontinues services. PAT uses development-centered parenting, family well-being, and community connections to reinforce this foundational curriculum.
  Arms: PAT as usual
Behavioral: Parents as Teachers (PAT) + Smart Parents — Added session to PAT following foundational visit 6. Smart Parents is comprised of 3 CSA specific prevention components: (1) healthy child sexual development, (2) communication about sexual concepts and sexual behaviors, and (3) safety strategies (including online safety.
  Delivered in one session (~60 min). Parents return to PAT as usual following this session.
  Arms: PAT + Smart Parents

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a parent-focused child sexual abuse prevention program (Smart Parents) delivered to parents enrolled in a parent education program (Parents as Teachers; PAT). The main questions the trial aims to answer are:

1. Does PAT + Smart Parents improve parents' CSA-related awareness and protective behaviors compared to PAT as usual?
2. Are potential gains maintained 12- and 24-months post intervention?
3. What parent-, provider-, and organizational-level factors hold promise for future dissemination and implementation efforts?

DETAILED DESCRIPTION:
To expand the empirical evidence for the effectiveness of Smart Parents and to explore the implementation factors that might promote or hinder adoption, fidelity, and scalability, the proposed study uses a type 2 hybrid effectiveness-implementation design. Designed to efficiently bridge the research to practice gap, the type 2 hybrid design tests the effectiveness of an intervention while concurrently exploring the viability of an explicit implementation strategy in a real world setting. To determine effectiveness (Aims 1 & 2), the investigators will conduct a pragmatic, quasi-experimental, stepped wedge cluster randomized trial (SW-CRT; N = 400) of CSA-related awareness (i.e., knowledge and attitudes about CSA and CSA prevention) and intention to use CSA protective behaviors for parents receiving Smart Parents when added to PAT (PAT+Smart Parents) compared to parents receiving PAT treatment as usual (PAT-TAU; Aim 1). The investigators will follow-up participating parents in both conditions at 12- and 24-months to determine retention of awareness (i.e., knowledge and attitudes) and actual use of protective behaviors (Aim 2).

A variation of a crossover experimental design, the SW-CRT is a pragmatic experimental design wherein randomized clusters sequentially transition from control to intervention until all clusters are exposed to the intervention. Once introduced to a cluster, the intervention is never removed. Facilitated by PAT National, 25 PAT sites will be recruited at the start of the study period. Sites will then be randomized into 1 of 5 clustered sequences (or steps) each containing 5 sites (or clusters). At the time on randomization, providers at all sites will begin recruiting eligible parents for participation in research and parents will begin the data collection protocols. At the point of the wedge, sites will be trained to deliver Smart Parents and will transition from control (PAT+TAU) to intervention (PAT+Smart Parents) conditions, the timing of which will be determined by the randomized step assignment.

ELIGIBILITY:
Inclusion Criteria:

* One parent per household that is currently enrolled in PAT qualified to receive bi-weekly visits;
* English or Spanish speaking;
* Has at least one child at home over 12-mo;
* Only newly enrolled parents (i.e., parents who have not received more than 3 of the PAT foundational sessions).

Exclusion Criteria:

* Not currently enrolled in PAT;
* Not English or Spanish speaking;
* Does not have a child over 12-mo old;
* Previously enrolled in PAT (i.e., parents who have received more than 3 of the PAT foundational sessions)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Sexual Abuse Knowledge | Baseline (T0)
  The Assessment of SmartParents Knowledge will be used to evaluate (a) CSA knowledge, norms, and attitudes (e.g., items regarding the degree to which parents endorsed accurate facts about CSA, the role of a parent in CSA prevention, and what is appropriate to discuss with children), and (b) intention to use CSA prevention related behaviors (e.g., items regarding identifying signs of CSA, talking to children and other adults about CSA prevention, and knowing how to respond appropriately if CSA is suspected).
Assessment of Sexual Abuse Knowledge | Up to 4 months (Post Session 6) (T1)
  The Assessment of SmartParents Knowledge will be used to evaluate (a) CSA knowledge, norms, and attitudes (e.g., items regarding the degree to which parents endorsed accurate facts about CSA, the role of a parent in CSA prevention, and what is appropriate to discuss with children), and (b) intention to use CSA prevention related behaviors (e.g., items regarding identifying signs of CSA, talking to children and other adults about CSA prevention, and knowing how to respond appropriately if CSA is suspected).
Assessment of Sexual Abuse Knowledge | 12-month assessment (T2)
  The Assessment of SmartParents Knowledge will be used to evaluate (a) CSA knowledge, norms, and attitudes (e.g., items regarding the degree to which parents endorsed accurate facts about CSA, the role of a parent in CSA prevention, and what is appropriate to discuss with children), and (b) intention to use CSA prevention related behaviors (e.g., items regarding identifying signs of CSA, talking to children and other adults about CSA prevention, and knowing how to respond appropriately if CSA is suspected).
Assessment of Sexual Abuse Knowledge | 24-month assessment (T3)
  The Assessment of SmartParents Knowledge will be used to evaluate (a) CSA knowledge, norms, and attitudes (e.g., items regarding the degree to which parents endorsed accurate facts about CSA, the role of a parent in CSA prevention, and what is appropriate to discuss with children), and (b) intention to use CSA prevention related behaviors (e.g., items regarding identifying signs of CSA, talking to children and other adults about CSA prevention, and knowing how to respond appropriately if CSA is suspected).
Parental Use of Behavioral Strategies Interview | 12-month assessment (T2)
  The Parental Use of Behavioral Strategies Interview (PUBSI) is a project created semi-structured behavioral interview deeply assess the use of behavior strategies at four levels: (1) community-level intentions, awareness, and behaviors; (2) personal environment; (3) personal actions/behaviors; and (4) personal behaviors. In addition to parents' reports of behaviors across the four levels, parents rate (on a scale of 1 to 5) their confidence in their ability to engage in each behavior as well as as their success in communicating with others about the various CSA related topics assessed.
Parental Use of Behavioral Strategies Interview | 24-month assessment (T3)
  The Parental Use of Behavioral Strategies Interview (PUBSI) is a project created semi-structured behavioral interview deeply assess the use of behavior strategies at four levels: (1) community-level intentions, awareness, and behaviors; (2) personal environment; (3) personal actions/behaviors; and (4) personal behaviors. In addition to parents' reports of behaviors across the four levels, parents rate (on a scale of 1 to 5) their confidence in their ability to engage in each behavior as well as as their success in communicating with others about the various CSA related topics assessed.
Preventive Behaviors Questionnaire | Baseline (T0)
  A 10-item instrument designed to assess the frequency with which parents perform protective behaviors within the past month (e.g., "Told my child never to keep secrets about touching" or "Talked to my relatives about my child's personal safety rules."). This quantitative assessment of behaviors will complement the PUBSI.
Preventive Behaviors Questionnaire | Up to 4 months (Post Session 6) (T1)
  A 10-item instrument designed to assess the frequency with which parents perform protective behaviors within the past month (e.g., "Told my child never to keep secrets about touching" or "Talked to my relatives about my child's personal safety rules."). This quantitative assessment of behaviors will complement the PUBSI.
Preventive Behaviors Questionnaire | 12-month assessment (T2)
  A 10-item instrument designed to assess the frequency with which parents perform protective behaviors within the past month (e.g., "Told my child never to keep secrets about touching" or "Talked to my relatives about my child's personal safety rules."). This quantitative assessment of behaviors will complement the PUBSI.
Preventive Behaviors Questionnaire | 24-month assessment (T3)
  A 10-item instrument designed to assess the frequency with which parents perform protective behaviors within the past month (e.g., "Told my child never to keep secrets about touching" or "Talked to my relatives about my child's personal safety rules."). This quantitative assessment of behaviors will complement the PUBSI.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, School of Global Public Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided